CLINICAL TRIAL: NCT03746106
Title: The Effect of SLC19A3 Inhibition on the Pharmacokinetics of Thiamine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tufts University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 13060; 5R01DK108722-02 (NIH)
Record Dates: First submitted 2018-11-08; First posted 2018-11-19 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Vitamin B1 Deficiency; Thiamine Deficiency
Keywords: Drug-induced vitamin deficiency
MeSH Terms: conditions — Beriberi; Thiamine Deficiency | interventions — Trimethoprim; Thymidine Monophosphate; Metformin; Thiamine

STUDY DESIGN:
Intervention Model Description: Part 1: Three-arm randomized crossover study design Part 2: Two-arm randomized crossover study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Thiamine only (Active Comparator): 5mg thiamine tablet by mouth. This arm will be included in both Parts 1 and 2 of the study.
  Interventions: Dietary Supplement: Vitamin B1
- Trimethporim + thiamine combination (Experimental): 5mg thiamine tablet and 300mg trimethoprim tablet by mouth. This arm will be included in both Parts 1 and 2 of the study.
  Interventions: Drug: Trimethoprim; Dietary Supplement: Vitamin B1
- Metformin + thiamine combination (Experimental): 5mg thiamine tablet and 1000mg metformin tablet by mouth. This arm will be included in only Part 1 of the study.
  Interventions: Drug: Metformin; Dietary Supplement: Vitamin B1

INTERVENTIONS:
Drug: Trimethoprim — 300mg of trimethoprim will be given in combination with 5mg thiamine and compared to 5mg thiamine only for both Parts 1 and 2 of the study.
  Other Names: Primsol
  Arms: Trimethporim + thiamine combination
Drug: Metformin — 1000mg of metformin will be given in combination with 5mg thiamine and compared to 5mg thiamine only in Part 1 of the study.
  Other Names: Glucophage
  Arms: Metformin + thiamine combination
Dietary Supplement: Vitamin B1 — 5mg of thiamine will be given alone and in combination for both Parts 1 and 2 of the study.
  Other Names: Thiamine

SUMMARY:
In Part 1, subjects will be administered thiamine, thiamine with metformin, and thiamine with trimethoprim. Part 2 will expand on Part 1 and subjects will be administered thiamine and thiamine with trimethoprim. The goal is to determine whether taking a drug and a vitamin together affects the body's ability to absorb, distribute, and eliminate thiamine (Vitamin B1).

DETAILED DESCRIPTION:
Thiamine is an essential vitamin meaning humans must consume thiamine from their diet in order to stay healthy. Low thiamine levels can lead to adverse events. Thiamine is absorbed in the intestine by a transporter protein. This is made by the SLC19A3 gene. The SLC19A3 gene provides instructions for making the thiamine transporter protein, which moves thiamine into cells. Certain drugs, like metformin and trimethoprim, have been shown to interrupt function of the SLC19A3 gene.

Metformin is a first-line therapy for patients with Type 2 diabetes and is associated with improvements in diabetic complications. Trimethoprim is an anti-bacterial drug that is often prescribed to treat infections such as urinary tract infections. At different phases of this study, participants will be administered thiamine, thiamine with metformin, and/or thiamine with trimethoprim to determine whether taking a drug and a vitamin together affects the body's ability to absorb, distribute, and eliminate thiamine. The levels of thiamine in the participants' blood and urine will be measured before and after taking thiamine or thiamine in combination with metformin and/or trimethoprim.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18-65 years old.
2. Eats a wide variety of food and willing to consume study diet (i.e. not on a specific diet such as Atkins, Fodmap, etc.).
3. Written informed consent obtained from the subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Subjects who are pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
2. Self-reported severe food allergies or diet restrictions (vegans, vegetarians, Atkins, Fodmap, etc.) that would prevent consumption of study diets.
3. Subjects with extreme obesity (BMI > 35).
4. Subjects who are smokers or have smoked in the past year and/or have smoked or ingested THC/marijuana in the past week, or who are unwilling to comply with a 1-week washout.
5. Subjects with any disease affecting or impairing the function of the liver, kidney or heart.
6. Subjects with moderate to severe hypertension.
7. Subjects with diabetes mellitus, hyperthyroidism, hypothyroidism, cardiovascular disease, glaucoma.
8. Subjects with gastrointestinal disease, gastrointestinal disorder, or gastrointestinal surgery.
9. Subjects with known infection with HIV, Hepatitis B (HBsAg) or Hepatitis C (no laboratory diagnostics concerning these diseases will be performed within the present study. Volunteers who are cured of past HepC infection are eligible to participate with doctor's approval letter).
10. Alcohol use on average > 2 servings/day or > 14 servings/wk (Serving size: 12oz beer/4oz wine/2oz hard liquor) or self-reported binge drinking.
11. Subjects that are on vitamin B supplements or multi-vitamins or who have taken vitamin B supplements or multi-vitamins in the past 30 days, or are not willing to comply with a 30-day washout of vitamin B supplements.
12. Subjects with possible folate deficiency.
13. Subjects taking any other clinically significant drugs as judged by the investigator.
14. Subjects with a condition, disease, or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
15. Female subjects undergoing treatment for infertility or hormone replacement therapy (Volunteers using hormonal birth control will not be excluded).
16. Subjects who have taken antimalarials in the past 60 days.
17. Participating in another research study while participating in this research study.
18. Non-English speaking
19. Subjects with abnormal laboratory results at screening as judged by the investigator or study physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Giacomini, Principal Investigator — University of California, San Francisco; Andrew S Greenberg, Principal Investigator — Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 subjects were randomized into one of two arms; each arm had two cycles (which were separated by a washout period of 5-14 days), and each cycle was three days in duration. During the Cycle 1, subjects were administered either a) 5 mg thiamine (n = 4) or b) 5 mg thiamine and 300 mg trimethoprim with 500 mL of water (n = 3). And during the Cycle 2, patients receive the other treatment.
Groups:
- Thiamine Alone, Then Thiamine Co-administered With Trimethoprim: One day prior to each study visit, participants arrived to collect three thiamine-deficient meals. They were instructed to consume these meals throughout the day, abstaining from other food intake. After an overnight fast, participants returned for their scheduled visit. On the first visit, they received 5 mg thiamine in 500 mL of water. Following a 5-14 day washout period, they repeated the process, this time receiving a combination of 5 mg thiamine and 300 mg trimethoprim with 500 mL of water.
- Thiamine Co-administered With Trimethoprim, Then Thiamine Alone: One day prior to each study visit, participants arrived to collect three thiamine-deficient meals. They were instructed to consume these meals throughout the day, abstaining from other food intake. After an overnight fast, participants returned for their scheduled visit. On the first visit, they received a combination of 5 mg thiamine and 300 mg trimethoprim with 500 mL of water. Following a 5-14 day washout period, they repeated the process, this time receiving a 5 mg thiamine in 500 mL of water.
Period: Cycle 1
Arm/Group | Thiamine Alone, Then Thiamine Co-administered With Trimethoprim | Thiamine Co-administered With Trimethoprim, Then Thiamine Alone
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0
Period: Cycle 2
Arm/Group | Thiamine Alone, Then Thiamine Co-administered With Trimethoprim | Thiamine Co-administered With Trimethoprim, Then Thiamine Alone
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Thiamine Alone, Thiamine Co-administered With Trimethoprim: Subjects were randomized into one of two arms; each arm had two cycles (which were separated by a washout period of 5-14 days), and each cycle was three days in duration. During the Cycle 1, subjects were administered either a) 5 mg thiamine (n = 4) or b) 5 mg thiamine and 300 mg trimethoprim with 500 mL of water (n = 3). And during the Cycle 2, patients receive the other treatment.
Arm/Group | Thiamine Alone, Thiamine Co-administered With Trimethoprim
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 2
Weight [Mean (Standard Deviation); unit: kg] | 76 (16)
Height [Mean (Standard Deviation); unit: cm] | 170 (7.3)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.4 (4.6)
Baseline Thiamine (Thiamine arm) [Mean (Standard Deviation); unit: nM] | 12.3 (24.0)
Baseline Thiamine (Trimethoprim + Thiamine arm) [Mean (Standard Deviation); unit: nM] | 4.5 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration (Cmax) of Thiamine in Plasma Between the Combination Arm(s) and Single Agent Arm
Description: Plasma samples were collected at pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, and 24 hours post-dose for each cycle. Cmax is determined by taking blood samples at various time points after drug administration and analyzing the thiamine concentration in plasma.
Time Frame: The highest concentration of a thiamine observed in the blood plasma after drug administration
Measure: Mean (Standard Deviation); unit: nM
Groups:
- Thiamine Alone: Participants who received 5 mg thiamine in 500 mL of water in either the first or second cycle of the study.
- Thiamine Co-administered With Trimethoprim: Participants who received a combination of 5 mg thiamine and 300 mg trimethoprim with 500 mL of water in either the first or second cycle of the study.
Arm/Group | Thiamine Alone | Thiamine Co-administered With Trimethoprim
Number analyzed (Participants) | 7 | 7
nM | 15 (9.5) | 32 (22)

2. Primary Outcome: Area Under the Curve From 0 to 24 (AUC0-24)Hours of Thiamine in Plasma Between the Combination Arm(s) and Single Agent Arm
Description: Plasma samples were collected at pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, and 24 hours post-dose for each cycle. AUC0-24 (Area Under the Curve from 0 to 24 hours) is a pharmacokinetic (PK) parameter that represents the total drug exposure in the body over a 24-hour period. It is calculated as the area under the plasma thiamine concentration vs. time curve (from time zero to 24 hours after drug administration).
Time Frame: Plasma samples were collected at pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, and 24 hours post-dose for each cycle.
Measure: Mean (Standard Deviation); unit: nM*hr
Arm/Group | Thiamine Alone | Thiamine Co-administered With Trimethoprim
Number analyzed (Participants) | 7 | 7
nM*hr | 50 (30) | 189 (138)

ADVERSE EVENTS:
Time Frame: Two cycles (which were separated by a washout period of 5-14 days) and each cycle was three days in duration.
Description: The safty population included all participants who received the drug. The National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 should be used to assess and grade adverse event severity, including laboratory abnormalities judged to be clinically significant.
Arm/Group | Thiamine Alone | Thiamine Co-administered With Trimethoprim
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (5):
  • Study Protocol and Statistical Analysis Plan (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT03746106/Prot_SAP_000.pdf
  • Informed Consent Form: Main ICF Part 2 (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT03746106/ICF_001.pdf
  • Informed Consent Form: Screening ICF Part 2 (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT03746106/ICF_002.pdf
  • Informed Consent Form: Main ICF (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT03746106/ICF_003.pdf
  • Informed Consent Form: Screening ICF (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT03746106/ICF_004.pdf